CLINICAL TRIAL: NCT07252141
Title: Association Between the Expression Levels of MicroRNA-101-3p and Autotaxin in Serum of Systemic Lupus Erythematosus Patients
Brief Title: miR-101-3p and Autotaxin in SLE Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Eman Mohamed Shawky (Other)
Responsible Party: Sponsor-Investigator, Eman Mohamed Shawky, Lecturer of Rheumatology and Rehabilitation, Faculty of Medicine, Assiut University, Assiut University
Organization: Assiut University (Other)
Other Study IDs: IRB.no: 04-2025-300546
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Forty patients diagnosed with systemic lupus erythematosus and Forty healthy control group: SLE Patients
  Group/Cohort Description: Forty patients diagnosed with systemic lupus erythematosus according to the 2012 Systemic Lupus International Collaborating Clinics (SLICC) classification criteria. Clinical and laboratory data, including disease activity indices (SLEDAI-2K and SDI), will be collected. Serum samples will be analyzed for miR-101-3p expression (qRT-PCR) and Autotaxin levels (ELISA).
  - Group/Cohort 2
  Group/Cohort Label:
  Healthy Controls
  Group/Cohort Description:
  Forty age- and sex-matched healthy individuals without autoimmune, infectious, or chronic inflammatory diseases. Blood samples will be collected for serum miR-101-3p and Autotaxin assessment using the same methods applied to the patient group.

SUMMARY:
Systemic lupus erythematosus (SLE) is a complex autoimmune disease affecting multiple organs and characterized by heterogeneous clinical manifestations. This case-control study aims to assess the association between serum expression levels of MicroRNA-101-3p and Autotaxin (ATX) in SLE patients compared with healthy controls. The hypothesis is that dysregulation of miR-101-3p and ATX contributes to SLE pathogenesis and may serve as potential non-invasive biomarkers for disease activity and prognosis.

DETAILED DESCRIPTION:
This descriptive case-control study will enroll 40 SLE patients fulfilling the 2012 Systemic Lupus International Collaborating Clinics (SLICC) classification criteria and 40 age- and sex-matched healthy individuals. Demographic, clinical, and laboratory data will be collected, including disease duration, activity indices (SLEDAI-2K), and damage index (SDI). Blood samples will be taken for biochemical and molecular analyses. Serum miR-101-3p expression will be quantified by qRT-PCR, while Autotaxin and IL-6 levels will be measured by ELISA. Statistical correlations between these biomarkers and clinical variables will be evaluated. The study aims to identify diagnostic and prognostic biomarkers that may guide future therapeutic targets in SLE.

ELIGIBILITY:
Inclusion Criteria:

* Study Population: Adult patients diagnosed with systemic lupus erythematosus and healthy matched controls.

Inclusion Criteria:

* - Age ≥ 18 years
* Diagnosis of SLE according to 2012 SLICC criteria
* Willingness to participate and provide informed consent

Exclusion Criteria: Age < 18 years

* Pregnancy or lactation
* Active infections or malignancy
* Co-existing autoimmune diseases
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include 40 patients diagnosed with systemic lupus erythematosus (SLE) according to the 2012 Systemic Lupus International Collaborating Clinics (SLICC) classification criteria and 40 age- and sex-matched healthy controls. Patients will be recruited from the Rheumatology and Rehabilitation Department and Internal Medicine Department (Rheumatology Unit) at Assiut University Hospitals, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Serum levels of miR-101-3p and Autotaxin in SLE patients versus healthy controls | 6 months (expected)
  To determine the difference in serum expression levels of miR-101-3p and Autotaxin between patients with systemic lupus erythematosus (SLE) and age- and sex-matched healthy controls using qRT-PCR and ELISA.

SECONDARY OUTCOMES:
Correlation between miR-101-3p and Autotaxin levels | 6 monthes expected
  To evaluate the relationship between serum miR-101-3p and Autotaxin concentrations in SLE patients.